CLINICAL TRIAL: NCT02069834
Title: Dolutegravir + Rilpivirine Switch Study (DORISS): Pilot and Noninferiority Trial Comparing Dolutegravir + Rilpivirine vs. Continued HAART (Highly Active Antiretroviral Therapy) in Patients With Plasma HIV RNA ≤ 50 Copies/mL for at Least 2 Years
Brief Title: Dolutegravir + Rilpivirine Switch Study (DORISS)
Acronym: DORISS
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: One of the both Funder partners decided to stop the study before the initiation : thus no product provided and no funding to realize the study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0322; 2013-003344-23 (EudraCT Number)
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infection; HAART-treated; Virologically Controlled
Keywords: Dolutegravir; Rilpivirine; PI- and NRTI- sparing ART regimen; switch study
MeSH Terms: conditions — HIV Infections | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (intervention) (Experimental): Dolutegravir 50 mg/d + Rilpivirine 25 mg/d qd orally (intake during a meal)
  Interventions: Drug: Arm 1 (intervention)
- Arm 2 (control) (Active Comparator): Continuation of existing HAART at the time of randomization
  Interventions: Drug: Arm 2 (control)

INTERVENTIONS:
Drug: Arm 1 (intervention) — Dolutegravir 50 mg/j + Rilpivirine 25 mg/j qd orally (intake during meal)
  Arms: Arm 1 (intervention)
Drug: Arm 2 (control) — Continuation of existing HAART at the time of randomization
  Arms: Arm 2 (control)

SUMMARY:
The primary objective of the study is to evaluate the capacity of Dolutegravir + Rilpivirine vs. continued triple combination HAART to maintain plasma HIV RNA ≤ 50 copies/ml throughout 24 weeks in patients with plasma HIV RNA ≤ 50 copies/mL for at least 2 years under conventional HAART (2 NNRTI + 3rd agent).

The main secondary objectives are the following:

* % of virologic success (plasma viral load ≤ 50 copies/mL) at W24 and W48
* % of patients who maintain a plasma viral load ≤ 50 copies / ml from D0 to W48
* % of virological failure defined by two consecutive plasma viral load > 50 copies/mL
* Profile of genotypic resistance in case of virological failure.

The trial will be conducted according to the design below, in 3 steps:

* Step 1: enrollment of 80 patients (40 in each arm)
* Step 2: enrollment on hold until W16 data from the 40 patients enrolled in the intervention arm have been analyzed.
* Step 3: resumption and completion of enrollment if conditions for resuming enrollment at the end of step 2 are fulfilled, i.e. if the percentage of patients randomized to the intervention arm who have a plasma viral load ≤ 50 copies/mL from D0 to W16 is significantly > 70%, which translates in a maximum of 6 virologic failures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV-1 infection
* Treatment with suppressive triple HAART (2 NRTI + either 1 PI/r, or 1 NNRTI, or INI), unchanged for > 6 months, Intra-class substitution within past 6 months is not considered as a treatment change.
* Plasma HIV-RNA ≤ 50 copies/mL for > 2 years
* CD4 cell count > 350/mm3 for > 6 months
* No prior virologic failure under an NNRTI-containing or an INSTI-containing ART regimen
* No NNRTI mutation on pre-ART genotype (if no pre-ART genotype available: no NNRTI mutation on DNA genotype at screening) among the following: K101E/P, E138A/G/K/Q/R/S, V179L, Y181C/I/V, Y188L, H221Y, M230I/L/V, L100I + K103N/S, L100I +K103R +V179D.
* No mutation (either on pre-ART genotype or on DNA genotype at screening) among the following: T66K, G118R, V151L, S153F/Y, R263K, T66K + L74M, E92Q + N155H, Q148R +N155H, Q148H/K/R with at least one mutation of L74I or E138A/K/T or G140A/C/S
* Negative HBs Ag
* Informed consent form signed by patient and investigator
* A specific consent for the pharmacokinetic substudy will be signed by the 10 patients of the pilot phase of the trial who will be randomized to the Dolutegravir + Rilpivirine arm and will volunteer for this PK study
* Patient covered with health insurance
* Effective contraception

Exclusion Criteria:

* HIV-2 infection
* Dialysis or severe renal failure (creatinine clearance < 30 ml/min)
* History of decompensated liver disease
* History of HIV-associated neurocognitive disorders
* AST or ALT > 5 x ULN
* Positive HBc Ac and negative HBs Ac
* Patient receiving a proton pump inhibitor that cannot be switched to another anti-secretory drug
* Current pregnancy or breastfeeding
* Patient involved in another research that precludes enrolment in another trial
* Patient under guardianship, or deprived of liberty by a court or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Pilot phase: Percentage of patients with plasma viral load ≤ 50 copies HIV-RNA/ml from D0 (Day 0) to W16 (Week 16) | Week 16
Non-inferiority phase: Percentage of patients with plasma HIV RNA maintained ≤ 50 copies/mL throughout 24 weeks | Week 24

SECONDARY OUTCOMES:
Percentage of patients with plasma viral load ≤50 HIV RNA copies/mL at Week 24 and Week 48 | Week 48
Percentage of patients with plasma viral load ≤50 HIV RNA copies/mL from Day 0 to Week 48 | Week 48
Percentage of virologic failure, defined as 2 consecutive plasma HIV RNA > 50 copies/mL | Week 48
Measure of the profile of genotypic resistance in plasma in case of virologic failure | Week 48
Percentage of patients who discontinued or changed the strategy of the study | Week 48
Measure of the HIV-DNA between day 0 and week 48 | W48
  Evolution of the HIV-DNA between Day 0 and week 48
Measure of CD4 lymphocytes at week 24 compared to day 0 | Week 24
  Evolution of CD4 lymphocytes (average) at Week 24 compared to Day 0
Measure of CD4 lymphocytes at Week 48 compared to Day 0 | Week 48
  Evolution of CD4 lymphocytes (average) at Week 48 compared to Day0
Number of patients with adverse events of grade 2 to 4 | Week 48
  Adverse events : incidence, grade and relation to study medication of all adverse events, of grade 2 to 4 events
Measure of changes in serum plasma lipid parameters at week 24 compared to Day 0 | Week 24
  Mean changes in serum plasma lipid parameters at Week 24 compared to Day 0
Measure of changes in serum lipid parameters at week 48 to Day 0 | Week 48
  Mean changes in serum plasma lipid parameters at Week 48 compared to Day 0
Measure of changes in fat mass distribution at week 24 compared to Day 0 | Week 24
  Changes in fat mass distribution at Week 24 compared to Day 0
Measure of changes in fat mass distribution at Week 48 compared to Day 0 | Week 48
  Changes in fat mass distribution at Week 48 compared to Day 0
Measure of adherence to treatment at Week 24 compared to Day 0 | Week 24
  Evolution of adherence to treatment at Week 24 compared to Day 0 assessed by a validated questionnaire
Measure of adherence to treatment at Week 48 compared to Day 0 | Week 48
  Evolution of adherence to treatment at Week 48 compared to Day 0 assessed by a validated questionnaire
Measure of patient satisfaction for their treatment at Day 0 | Day 0
  Assessment of patient satisfaction for their treatment at D0 by questionnaire
Measure of patient satisfaction for their treatment at Week 24 | Week 24
  Assessment of patient satisfaction for their treatment at Week 24 by questionnaire
Measure of patient satisfaction for their treatment at Week 48 | Week 48
  Assessment of patient satisfaction for their treatment at Week 48 by questionnaire
Measure of changes in plasma biomarkers of inflammation (hs-CRP and IL-6) and immune activation (sCD14 , MCP -1, IP10 ) at Week 24 compared to Day 0 . | Week 24
  Changes in plasma biomarkers of inflammation (hs-CRP and IL-6) and immune activation (sCD14 , MCP -1, IP10 ) at Week 24 compared to Day 0 .
Measure of changes in plasma biomarkers of inflammation (hs-CRP and IL-6) and immune activation (sCD14 , MCP -1, IP10 ) at Week 48 compared to Day 0 . | Week 48
  Changes in plasma biomarkers of inflammation (hs-CRP and IL-6) and immune activation (sCD14 , MCP -1, IP10 ) at Week 48 compared to Day 0 .
Measure of plasma concentrations of Dolutegravir and Rilpivirine measured at Week 4 | Week 4
  Analysis PK (PharmacoKinetic) / PD (Pharmaodynamic) of plasma concentrations of Dolutegravir and Rilpivirine measured at Week 4
Measure of plasma concentrations of Dolutegravir and Rilpivirine measured at Week 24 | Week 24
  Analysis PK / PD of plasma concentrations of Dolutegravir and Rilpivirine measured at Week 24
Measure of the profile of genotypic resistance in plasma in case of virologic failure | Week 24
Percentage of virologic failure, defined as 2 consecutive plasma HIV RNA > 50 copies/mL | Week 24

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - CHU Guadeloupe, Point-a-pitre, Guadeloupe
  - CHU de Fort de France, Fort de France, Martinique
  - Chu Jean Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital Jean Verdier, Bondy
  - CHU de Bordeaux, Bordeaux
  - CHU de DIJON, Dijon
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - CHU Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Perpetuel Secours, Levallois-Perret
  - CHU de Nantes, Nantes
  - CHU Hôtel Dieu Paris, Paris
  - Hôpital La Pitié Salpêtrière, Paris
  - Hôpital Necker - enfants Malades, Paris
  - Hôpital Saint Louis, Paris
  - CHU BICHAT - Claude Bernard, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - CH Delafontaine, Saint-Denis
  - CHU Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - CHU Toulouse, Toulouse
  - CHRU de Tours, Tours
  - CHU de Nancy, Vandœuvre-lès-Nancy